CLINICAL TRIAL: NCT04194489
Title: Feasibility Trial of the FMF Connect Mobile Health Intervention
Brief Title: Trial of the Families Moving Forward (FMF) Connect Mobile Health Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christie Petrenko, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4433; U01AA026104 (NIH)
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMF Connect Intervention (Experimental)
  Interventions: Other: FMF Connect

INTERVENTIONS:
Other: FMF Connect — The FMF Connect intervention includes cloud infrastructure and an innovative, multilayered mobile app. It incorporates tailored content for parents/caregivers of children (ages 3-12) with FASD or PAE. The app integrates five main components: 1) Dashboard; 2) Learning Modules; 3) Family Forum; 4) Library; and 5) Notebook. Weekly emails are also sent to support motivational engagement.

SUMMARY:
The purpose of this study is to test a new smartphone "app" for parents/caregivers of children with fetal alcohol spectrum disorder (FASD). The app is called Families Moving Forward (FMF) Connect. The goal of the app is to provide parents/caregivers with useful information to help manage their children's condition and obtain peer support.

ELIGIBILITY:
Inclusion Criteria:

* Biological parent or other primary caregiver (e.g., foster or adoptive parent, relative, legal guardian) of a child with FASD or prenatal alcohol exposure (PAE)
* The parent/caregiver must be at least 18 years old
* The child must between the ages of 3 and 12 years old
* The child has a diagnosis of FASD or has confirmed PAE
* The child has lived with the parent/caregiver for at least 4 months and is expected to remain in the home for at least 1 year
* The parent/caregiver lives in the United States
* The parent/caregiver has a smartphone with iOS or Android operating system

Exclusion Criteria:

* The parent/caregiver is not fluent in English (the FMF Connect app and pre-post measures are currently only available in English)
* There is another parent/caregiver of the same child or living in the home that is already enrolled in the study (couples are excluded to prevent dependence in the data)
* The family has previously received or is currently receiving the therapist-led Families Moving Forward (FMF) Program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is deposited quarterly into the Collaborative Initiative on Fetal Alcohol Spectrum Disorders central repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It will be available once the data is collected and will be available indefinitely.
URL: http://www.cifasd.org/data-sharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were asked to complete an eConsent and several screening questionnaires in REDCap. A total of 66 did not proceed to assignment to study arm for the following reasons: 24 did not meet eligibility criteria, 38 had incomplete data so eligibility was not able to be determined, 3 chose to wait for the subsequent RCT, and 1 was overlooked due to study team error.
Period: Overall Study
Arm/Group | FMF Connect Intervention
Started | 105
Completed Some or All Baseline Surveys | 85
Installed FMF Connect App | 67
Completed Some or All Follow-up Surveys | 52
Completed | 52
Not Completed | 53
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 48

BASELINE CHARACTERISTICS:
Population: A total of 105 participants were assigned to study arm. 5 withdrew from the study. Demographic data was collected during eligibility screening and reflects all 100 participants. A total of 85 participants started or completed baseline surveys. 1 participant completed only some measures.
Arm/Group | FMF Connect Intervention
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.48 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 92
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100
Relationship to Child [Number; unit: participants] — A total of 8 participants belonged to multiple categories.
  participants
    Biological Parent | 3
    Adoptive Parent | 83
    Foster Parent | 7
    Grandparent | 7
    Other Relative | 8
Phone Operating System [Count of Participants; unit: Participants]
  Apple iOS | 62
  Android | 38
Child Age [Mean (Standard Deviation); unit: years] | 8.09 (2.62)
Child Sex at Birth [Count of Participants; unit: Participants]
  Male | 61
  Female | 39
Child Race [Count of Participants; unit: Participants]
  African American / Black | 6
  Asian | 2
  White | 59
  Native American / Alaska Native | 6
  Native Hawaiian / Pacific Islander | 1
  More Than One Race | 23
  Unknown | 3
Child Ethnicity [Count of Participants; unit: Participants]
  Hispanic / Latinx | 16
  Not Hispanic / Latinx | 80
  Unknown | 4
Eyberg Child Behavior Inventory - Intensity [Mean (Standard Deviation); unit: units on a scale] — Population: Data presented includes all of those with baseline data collection for this measure.
  units on a scale
    number analyzed (Participants) | 85
    (all) | 69.75 (8.94)
Parenting Sense of Competence Scale - Efficacy [Mean (Standard Deviation); unit: units on a scale] — Population: Data presented is only from participants who have complete data for this measure.
  units on a scale
    number analyzed (Participants) | 84
    (all) | 21.17 (5.48)
Parenting Sense of Competence Scale - Satisfaction [Mean (Standard Deviation); unit: units on a scale] — Population: Data presented includes only those participants who have complete data for this measure.
  units on a scale
    number analyzed (Participants) | 85
    (all) | 34.29 (6.43)
Family Needs Met Scale [Mean (Standard Deviation); unit: units on a scale] — Population: Data is presented for participants with complete data on this measure.
  units on a scale
    number analyzed (Participants) | 85
    (all) | 2.35 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Eyberg Child Behavior Inventory at Baseline and 3-Month Follow-Up
Description: The Eyberg Child Behavior Inventory measures the intensity of child behavior problems. Scores are presented as T-scores with a mean of 50 and a standard deviation of 10. A T-score of 60 or higher is considered clinically significant. Higher scores indicate more intense behavior problems. An effect size of 0.2 is small, 0.5 is medium and 0.8 is large.
Time Frame: baseline to 3-month follow-up
Population: Data was analyzed from participants with complete data on the measure from both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMF Connect Intervention
Number analyzed (Participants) | 52
score on a scale
  Baseline | 69.31 (9.29)
  Follow-up | 65.62 (7.81)
Statistical Analysis 1: Comparison: FMF Connect Intervention; Cohen's d effect size was calculated using baseline and follow-up means and standard deviations. An effect size of 0.2 is small, 0.5 is medium and 0.8 is large; Test type: Other — Effect size calculation; Cohen's d = 0.43

2. Primary Outcome: Parenting Sense of Competence - Satisfaction Sub-scale at Baseline and 3-Month Follow-up
Description: The Parenting sense of competence scale includes two sub-scales: 1) satisfaction and 2) efficacy. The satisfaction sub-scale reported here includes 9 items, rated on a scale from 1 ("strongly agree") to 6 ("strongly disagree"). Responses are summed, with possible sub-scale score range from 9 to 54 with higher scores indicating higher satisfaction in the parenting role. An effect size of 0.2 is small, 0.5 is medium and 0.8 is large.
Time Frame: baseline to 3-month follow-up
Population: Data was analyzed from participants with complete data on the measure from both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMF Connect Intervention
Number analyzed (Participants) | 52
score on a scale
  Baseline | 32.90 (6.18)
  Follow-up | 34.02 (7.18)
Statistical Analysis 1: Comparison: FMF Connect Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Other — Effect size; Cohen's d = 0.17

3. Primary Outcome: Parenting Sense of Competence - Efficacy Sub-scale Baseline to 3-Month Follow-up
Description: The Parenting sense of competence scale includes two sub-scales: 1) satisfaction and 2) efficacy. The efficacy sub-scale reported here measures how effective parents feel they are and includes 7 items, rated on a scale from 1 ("strongly agree") to 6 ("strongly disagree"). Responses are summed, with possible sub-scale score range from 7 to 42 with higher scores indicating lower feelings of efficacy. An effect size of 0.2 is small, 0.5 is medium and 0.8 is large.
Time Frame: baseline to 3-month follow-up
Population: Data was analyzed from participants with complete data on the measure from both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMF Connect Intervention
Number analyzed (Participants) | 52
score on a scale
  Baseline | 22.04 (6.01)
  Follow-up | 20.56 (4.80)
Statistical Analysis 1: Comparison: FMF Connect Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Other — Effect size calculation; Cohen's d = 0.27

4. Primary Outcome: Family Needs Questionnaire Baseline to 3-Month Follow-up
Description: The family needs questionnaire measures the degree to which family needs are met. The scale includes 20 items reflecting family needs that are rated on a scale from 0 to 4, with 0 being not applicable to 4 being met a great deal. The total score on this measure is created by averaging across all items. Total score ranges from 0-4. Higher scores reflect more needs being met. An effect size of 0.2 is small, 0.5 is medium and 0.8 is large.
Time Frame: baseline to 3-month follow-up
Population: Data was analyzed from participants with complete data on the measure from both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMF Connect Intervention
Number analyzed (Participants) | 52
score on a scale
  Baseline | 2.34 (0.71)
  Follow-up | 2.35 (0.57)
Statistical Analysis 1: Comparison: FMF Connect Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Other — Effect size calculation; Cohen's d = 0.02

5. Secondary Outcome: Participant Perception of Self-care Change Over Intervention Period Reported at 3-month Follow-up
Description: Participants are asked at follow-up to rate how much their self-care practices have changed over the last 3 months on a 5-point scale ranging from "A lot less self-care (1)" to "A lot more self-care (5)." A score of 3 equates to no change.
Time Frame: 3-month follow-up
Population: Data was analyzed from participants with complete data on the measure at the 3-month follow-up timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMF Connect Intervention
Number analyzed (Participants) | 52
score on a scale | 2.92 (1.22)

6. Secondary Outcome: Mean App Quality Score on Mobile App Rating Scale: User Version
Description: The mobile app rating scale includes a measure of users perception of app quality. There are 16 items contributing to this score, each rated on a scale from 1 to 5. Total app quality score is presented as a mean with range of 1 to 5, with higher scores reflecting greater perceived quality of the app. .
Time Frame: 3-month follow-up
Population: Data was analyzed from participants with complete data on the measure at the 3-month follow-up timepoint. Data was missing for 2 participants on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMF Connect Intervention
Number analyzed (Participants) | 50
score on a scale | 4.08 (0.47)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events in children with FASD or their caregivers could include aggression or violence towards others, maltreatment, self-harm or suicidality, or the need for inpatient hospitalization. However, these occurrences are unlikely to be a direct consequence of participation in the caregiver intervention or study. These were not systematically assessed but procedures were in place to assess risk and respond appropriately if they arose.
Arm/Group | FMF Connect Intervention
All-Cause Mortality (participants affected / at risk) | 0/105
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 0/105

LIMITATIONS AND CAVEATS:
This study was designed to assess intervention and trial feasibility rather than test efficacy. Effect sizes were calculate to estimate sensitive of selected measures to change and inform refinements prior to RCT. Also note, Android participants completed study procedures almost a year later than iOS due to COVID-19 pandemic-related project delays.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT04194489/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT04194489/ICF_001.pdf